CLINICAL TRIAL: NCT06704100
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Trial of Fosamprenavir-Sodium Alginate Administered Orally for 8 Weeks to Patients With Proton Pump Inhibitor Refractory Gastroesophageal Reflux Disease
Brief Title: Oral Fosamprenavir + Sodium Alginate for GERD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Nikki Johnston, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO000000000
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Refractory Gastroesophageal Reflux Disease; Gastroesophageal Reflux Disease
Keywords: PPI-refractory GERD; Proton pump inhibitor refractory gastroesophageal reflux disease; Fosamprenavir; Sodium Alginate; Fosamprenavir-Sodium Alginate; FOS-SA
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — fosamprenavir; Alginates; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Proof-of-Concept
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We have partnered with Froedtert Hospital's Investigative Drug Services (FH IDS) in order to randomize subjects to either treatment or placebo. Only FH IDS will have the key linking subjects to treatment groups, and the power to conduct an emergency un-blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Fosamprenavir-Sodium Alginate (FOS-SA) (Experimental): Eight weeks of:
  1400 mg FOS-SA BID: 15 ml oral solution containing 1400 mg fosamprenavir calcium and 24.5 mg sodium alginate administered BID, at least 1 hour before or 2 hours after the morning and evening meals, approximately 12 hours apart
  Interventions: Drug: Fosamprenavir Calcium & Sodium Alginate
- Oral Placebo (Placebo Comparator): Eight weeks of:
  15 ml oral solution containing 1,399 mg microcrystalline cellulose and 24.5 mg sodium alginate administered BID at least 1 hour before or 2 hours after the morning and evening meals, approximately 12 hours apart
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fosamprenavir Calcium & Sodium Alginate — 1400 mg FOS-SA BID: 15 ml oral solution containing 1400 mg fosamprenavir calcium and 24.5 mg sodium alginate administered BID
  Arms: Oral Fosamprenavir-Sodium Alginate (FOS-SA)
Other: Placebo — 15 ml oral solution containing 1,399 mg microcrystalline cellulose and 24.5 mg sodium alginate
  Other Names: Microcrystalline cellulose; Sodium Alginate
  Arms: Oral Placebo

SUMMARY:
The goal of this clinical trial is to learn if study drug Fosamprenavir-Sodium Alginate (FOS-SA) administered orally improves symptoms for Proton Pump Inhibitor (PPI)-refractory Gastro Esophageal Reflux Disease (GERD).

The main questions it aims to answer are:

1. Does FOS-SA significantly improve heartburn severity over the 8-week treatment period
2. Does FOS-SA significantly improve regurgitation frequency over the 8-week treatment period
3. Does FOS-SA significantly improve symptoms of persistent GERD over the 8-week treatment period

Researchers will compare FOS-SA to a placebo (a look-alike substance that contains no active drug) to see if FOS-SA works to treat PPI-refractory GERD.

Participants will:

1. Take FOS-SA or placebo every day BID (twice a day) for 8 weeks
2. Visit the Adult Translational Research Unit (ATRU) seven times for consenting, screening, and checkups and tests
3. Keep a daily diary of their symptoms of persistent GERD

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18-65 selected as candidate for anti-reflux surgery by study providers.
2. Patient has received, and continued having GERD symptoms during, standard-labeled dose, daily, PPI therapy for a minimum of 8 weeks before the Screening Visit.
3. Patient has a diagnosis of GERD with endoscopy and/or pH-metry test within the past two years demonstrating 1 or more of the following:

   1. Erosive esophagitis (Grade A or greater based on the Los Angeles classification of esophagitis; Appendix 3)
   2. Evidence of pathological acid reflux (pH < 4 for ≥ 4-6% off therapy or ≥ 1-4% on therapy) during a 24-hour time interval of pH testing
4. Patient reports heartburn severity (HS, Item #1 on mRESQ-eD) ≥ 3 (moderate) on at least 2 days and has an average HS of ≥ 2 (mild) during the last 7 days of the Pretreatment Period before Randomization.

Exclusion Criteria:

1. Patient is suspected of having, functional upper gastrointestinal disorders such as functional dyspepsia or functional heartburn diagnosed by the Rome IV criteria; Appendix 4.
2. Patient has endoscopically confirmed eosinophilic esophagitis (EE).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Weekly Heartburn Severity Score | Ten days of pre-screening and dailyfor 8 weeks.
  Based on questions 1 and 2 of mRESQ-eD. The percent change from baseline (i.e., Pretreatment) in heartburn severity as indicated by Weekly Heartburn Severity Score (WHSS) at Week 8 (end of Treatment Period). Weekly scoring averaged.
  [Minimum Value: 0, Maximum Value: 500, higher score= worse outcome]

SECONDARY OUTCOMES:
Weekly Regurgitation Frequency Score | Ten days of pre-screening and daily for 8 weeks.
  Based on questions 7 and 7 of mRESQ-eD. The percent change from baseline (i.e., Pretreatment) in regurgitation frequency as indicated by Weekly Regurgitation Frequency Score (WRFS) at Week 8. Weekly scoring averaged.
  [Minimum Value: 0, Maximum Value: 400, higher score= worse outcome]
Daily modified Reflux Symptom Questionnaire Electronic Diary (mRESQ-eD) | Ten days of pre-screening and daily for 8 weeks.
  The percent change from baseline (i.e., Pretreatment) in symptoms of persistent GERD as indicated by mRESQ-eD weekly total GERD score (WTGS) at Week 8. Weekly scoring averaged.
  [Minimum Value: 0, Maximum Value: 1850, higher score= worse outcome]

CONTACTS AND LOCATIONS:
Overall Officials: Nikki Johnston, PhD., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided